CLINICAL TRIAL: NCT06910358
Title: APOLLO: A Randomized, Double-Blind, Placebo-Controlled Study of Bitopertin to Evaluate the Efficacy, Safety, and Tolerability in Participants With Erythropoietic Protoporphyria (EPP) or X-Linked Protoporphyria (XLP)
Brief Title: Study of Bitopertin in Participants With EPP or XLP (APOLLO)
Acronym: APOLLO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DISC-1459-301; 2024-520407-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Erythropoietic Protoporphyria (EPP); X-Linked Protoporphyria (XLP)
Keywords: EPP; XLP; DISC-1459; RO4917838; porphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Protoporphyria, Erythropoietic, X-Linked Dominant; Porphyrias | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DISC-1459 oral dose (Experimental)
  Interventions: Drug: DISC-1459

INTERVENTIONS:
Drug: Placebo — Oral dose, once a day for 24 weeks
  Arms: Placebo
Drug: DISC-1459 — Oral dose, once a day for 24 weeks
  Other Names: Bitopertin; RO4917838
  Arms: DISC-1459 oral dose

SUMMARY:
The goal of this clinical trial is to learn if bitopertin works and is safe to treat EPP or XLP in participants 12 years or older. The main questions it aims to answer are:

* Whether bitopertin increases pain-free sunlight exposure after 6 months of treatment in participants with EPP or XLP.
* How PPIX concentration levels change from before bitopertin treatment to after 6 months of treatment.

Researchers will compare bitopertin to a placebo look-alike substance that contains no drug.

Participants will complete daily questionnaires and attend study visits for assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12 years or older at the time of study consent.
2. Diagnosis of EPP or XLP, based on medical history by ferrochelatase (FECH) or aminolevulinic acid synthase 2 (ALAS2) genotyping or by biochemical porphyrin analysis.
3. Minimum daily Sun Exposure Diary compliance ≥85% on Days -14 through Day -1, inclusive, during screening, and at least 1 successfully completed Sun Exposure Challenge (adults only, as this assessment is optional for adolescents) or historical recall of time to prodrome
4. Body weight ≥32 kg (ages 12 to <18 years), body mass index ≥18.5 kg/m2 (ages ≥18 years) at screening.
5. Washout of at least 2 months prior to screening of afamelanotide and dersimelagon, if applicable.
6. Aspartate aminotransferase and alanine transaminase <3× upper limit of normal (ULN)and total bilirubin <2× ULN (unless documented Gilbert syndrome) at screening. Albumin >lower limit of normal (LLN).
7. Willing to practice highly effective methods of birth control (both males who have partners of childbearing potential and females of childbearing potential during screening, while taking study drug, and for at least 30 days after the last dose of study drug).

Exclusion Criteria:

1. Major surgery within 8 weeks before screening or incomplete recovery from any previous surgery.
2. Other than EPP or XLP, an inherited intrinsic or extrinsic red cell disease associated with anemia.
3. Known hypersensitivity to any component of the study drug.
4. History of liver transplantation or anticipated need for liver transplantation.
5. History of alcohol dependence or excessive alcohol consumption, as assessed by the Investigator.
6. Active human immunodeficiency virus (HIV), active hepatitis B or C.
7. Other medical or psychiatric condition or laboratory finding not specifically noted above that, in the judgment of the Investigator or Sponsor, would put the participant at unacceptable risk or otherwise preclude the participant from participating in the study.
8. Condition or concomitant medication that would confound the ability to interpret clinical, clinical laboratory, or participant diary data, including a major psychiatric condition that has had an exacerbation or required hospitalization in the last 6 months.

   Treatment History:
9. Prior exposure to bitopertin.
10. Concurrent or planned treatment with afamelanotide or dersimelagon during the study period.
11. Treatment with opioids for any period >7 days in the 2 months prior to screening or anticipated to require opioid use for >7 days at any point during the study.
12. New treatment for anemia, including initiation of iron supplementation, within 1 month of screening.
13. Current or planned use of any drugs or herbal remedies known to be strong or moderate inhibitors or inducers of cytochrome P450 (CYP)3A4 enzymes for 28 days prior to the first dose and throughout the study.
14. Current or planned treatment with antipsychotic medication.

    Laboratory Exclusions:
15. Hemoglobin <10 g/dL at screening.

    Miscellaneous:
16. Participation in other interventional clinical studies within 30 days prior to screening.
17. If female, pregnant or breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Average monthly total time in sunlight on days without pain from a phototoxic reaction between 10:00 to 18:00 (10:00 AM to 6:00 PM) after 6 months (24 weeks) of treatment | 24 weeks
Percent change from baseline in whole-blood metal-free PPIX levels at 6 months | 24 weeks
Safety and tolerability, as assessed by adverse events (AEs) and laboratory results, over the 6-month treatment period | 24 weeks

SECONDARY OUTCOMES:
Occurrence of phototoxic reactions over the 6-month treatment period | 24 weeks
Cumulative total time in sunlight on days without pain from a phototoxic reaction between 10:00 to 18:00 (10:00 AM to 6:00 PM) over the 6-month (24-week) treatment period | 24 weeks
Change from baseline in 2-week average daily sunlight exposure time (minutes) to first prodromal symptom (eg, burning, tingling, itching, or stinging) associated with sunlight exposure between 1 hour post-sunrise and 1 hour pre-sunset at 6 months | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD, PhD, Study Director — Disc Medicine
Locations (23):
- United States (11):
  - Marvel Clinical Research, Huntington Beach, California
  - University of California San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - MetroBoston Clinical Partners, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mount Sinai Hospital, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Remington-Davis Clinical Research, Columbus, Ohio
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington, Seattle, Washington
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Royal Melbourne Hospital, Parkville, Victoria
- University of Alberta, Edmonton, Alberta, Canada
- France (2):
  - CHU de Nantes - Hôtel Dieu, Service de dermatologie, Nantes, France
  - Centre d'Investigation Clinique (CIC) Hôpital Bichat - Claude-Bernard, Paris, France
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Institute of Allergology, Berlin, Germany
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
- Erasmus MC, Rotterdam, The Netherlands, Netherlands
- Helse Bergen, Bergen, Norway, Norway
- Hospital Clinic de Barcelona, Barcelona, Spain, Spain
- Karolinska University Hospital, Stockholm, Sweden, Sweden
- Guy's and St Thomas' NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No